CLINICAL TRIAL: NCT00298922
Title: Phase II, Randomized, Double Blind, Placebo-Controlled Trial of Azithromycin in Patients With CF, Chronically Infected With Burkholderia Cepacia Complex
Brief Title: Azithromycin in Patients With CF, Infected With Burkholderia Cepacia Complex
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: Cystic Fibrosis Foundation (Other); Pfizer (Industry)
Responsible Party: Dr. Elizabeth Tullis, St. Michael's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AZ 0003; TULLIS04A0
Record Dates: First submitted 2006-03-02; First posted 2006-03-03 (Estimated); Last update posted 2009-07-31 (Estimated); Status verified 2009-07

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Burkholderia cepacia complex
MeSH Terms: conditions — Cystic Fibrosis | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Azithromycin (Active Comparator): participants taking 500 mg tablets orally thrice weekly for 24 weeks
  Interventions: Drug: Azithromycin
- Placebo (Placebo Comparator): Participants taking 500 mg tablets orally thrice weekly for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — 500 mg tablets orally thrice weekly for 24 weeks
  Arms: Azithromycin
Drug: Placebo — tablet orally thrice weekly for 24 weeks
  Arms: Placebo

SUMMARY:
Pulmonary infection with Burkholderia cepacia complex (BCC) in patients with CF is often associated with a more rapid decline in lung function. Because of the resistance of BCC to many antibiotics, treatment options are often limited. New therapies to improve outcomes for patients infected with BCC are needed.

However, because of the unpredictable nature of this pulmonary infection in CF, patients with BCC infection have been excluded from many CF therapeutic trials.

Recent published trials in the United States, Australia, and the United Kingdom have all demonstrated clinical benefits from prolonged administration of azithromycin in CF. In these trials, the vast majority of patients were chronically infected with Pseudomonas aeruginosa.

Patients with BCC were excluded from the US and UK trials, and only four patients with BCC infection were enrolled in the Australian trial. Thus, the effectiveness of azithromycin in CF patients infected with BCC is largely unknown and deserves further study.

The two main ways by which azithromycin is thought to help with the chronic lung infections seen in CF are by [a] reducing inflammation and [b] direct effects on the bacteria, in particular P. aeruginosa. BCC pulmonary infection in CF is often associated with a large inflammatory response similar to or more severe than P. aeruginosa infection. If azithromycin works mainly by an anti-inflammatory mechanism, it should also be helpful in CF patients infected with BCC.

Alternatively, azithromycin could have a direct effect on BCC as seen with P. aeruginosa as the two bacteria have many similarities.

DETAILED DESCRIPTION:
STUDY DESIGN

* Overview
* This is a single center, randomized, double-blinded, placebo-controlled 24 week trial of azithromycin in adults with CF chronically infected with BCC. The investigational therapy will be added to usual therapy in patients who are clinically stable at the time of enrollment. After 168 days, the study drug will be discontinued and participants will be evaluated at 196 days off of study drug for 28 days. At that visit, participants will be invited to continue in an open label observational study of azithromycin for 168 additional days. Thus, the duration of the study will be 52 weeks (364 days).
* Day 0- Day 168 on Study Drug (24 weeks)
* Day 169- Day 196 off Study Drug (4 weeks)
* Day 197 - Day 364 on OPEN label Azithromycin (24 weeks)
* Measuring primary and secondary endpoints
* Primary efficacy endpoint
* Primary efficacy endpoint will be the quantitative changes in lung function as measured by FEV1 in % predicted from baseline to completion of the 24 week treatment period. (refer to Appendix C for ATS guidelines).
* Primary safety endpoints
* Primary safety endpoints collected over the 24 week treatment period will be:

  * Adverse events such as gastrointestinal complaints, ototoxicity, tinnitus, hepatitis or leukopenia as determined by:

    (i) open ended questioning of study subjects at study visits (ii) laboratory tests for elevated liver function tests or hematologic abnormalities,
  * Changes in lung microbiology as determined by:[86] (i) Emergent B. cenocepacia (genomovar III) (ii) Emergent non-B. cenocepacia genomovars (iii) Emergent NTM[87] (iv) Emergent azithromycin resistant NTM (v) Emergent Aspergillus species (vi) Emergent MDRO - (S. maltophilia, A. xylosoxidans, or methicillin-resistant S. aureus) (vii) Emergent P. aeruginosa (viii) Emergent azithromycin resistant S. aureus
* Secondary efficacy endpoints
* Secondary efficacy endpoints will be:
* Quantitative changes in lung function as measured by change in relative percent change in FEV1 and FVC from baseline to completion of the 24 week treatment period.
* Quantitative change in FEV1 and FVC in liters in CF study subjects treated with azithromycin compared with those CF study subjects treated with placebo. FEV1 and FVC in liters will be measured according to ATS criteria
* The number of days until first administration of intravenous antibiotics and/or the use of oral tetracycline derivatives minocycline / doxycycline for seven or more days during the 24 week period.
* The number of pulmonary exacerbations as defined by need for treatment with intravenous or oral tetracycline derivative antibiotics for an increase in pulmonary symptoms during the 24 week period.
* The proportion of patients requiring intravenous antibiotics during the 24 week period.
* The number of days of treatment with intravenous antibiotics given during the 24 week period.
* The proportion of patients hospitalized.
* The number of hospital days as calculated by calendar days during the 24 week period.
* The proportion of patients requiring oral antibiotics during the 24 week period.
* The number of days of treatment with oral non-tetracycline derivative antibiotics given during the 24 week period.
* Changes in body weight from baseline to completion of the 24 week treatment period.
* Change in level of inflammation as measured by the change in serum CRP and ESR from baseline to the end of the 24 week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent and verbal assent as appropriate has been provided by the subject
* Ability to comply with medication use, study visits and study procedures as judged by the site Investigator
* Diagnosis of CF as defined by two or more clinical features of CF and a documented sweat chloride > 60 mEq/L by quantitative pilocarpine iontophoresis test or a genotype showing two well characterized disease causing mutations
* > 18 years of age
* Body weight > 40 kg
* BCC present in a sputum/throat culture > 1 year prior to screening and at screening
* FEV1 % predicted > 30% as calculated by the Knudsen reference equations
* Room air oximetry > 88% at rest
* Post-menarche females must be surgically sterile or using an effective form of contraception
* Predicted to live > 1 year and clinically stable at that time of enrollment as judged by the investigator.

Exclusion Criteria:

* History of chronic macrolide use, defined as regular macrolide antibiotic use within a three month period prior to enrollment in the study.
* AST or ALT > 2.5 times the upper limit of normal performed at the local laboratories on two occasions prior to randomization.
* Investigational drug use within 30 days of screening
* History of alcohol, illicit drug or medication abuse within 1 year of screening
* Use of intravenous antibiotics or oral antibiotics within 14 days of screening.
* Use of low dose oral antibiotics (e.g. macrolides, tetracycline, sulfa) for acne or other conditions within 30 days of screening
* Use of systemic corticosteroids (> 20 mg of prednisone per day) within 30 days of screening
* Initiation of TOBI®, high dose ibuprofen, or rhDNase within 60 days of screening
* History of lung transplantation or currently on lung transplant list
* History of allergy to a macrolide antibiotic
* AFB smear positive at screening suggesting current NTM infection.
* Positive serum pregnancy test at screening (to be performed on all post-menarche females)
* Absolute neutrophil count < 1000 performed at the local laboratories on two occasions prior to randomization
* Creatinine > 1.5 times normal performed at the local laboratories on two occasions prior to randomization.
* Chest x-ray changes or physical findings at screening that would compromise the safety of the patient or the quality of the study data
* Other major organ dysfunction

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2006-02; Primary Completion 2009-02 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Change in FEV1 in % predicted in CF study subjects treated with azithromycin compared with those CF study subjects treated with placebo. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Tullis, MD, Principal Investigator — University of Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada